CLINICAL TRIAL: NCT02093975
Title: Telemedical Solutions in Medical Emergencies, Advantages and Disadvantages for Patients, Healthcare Professionals, and Healthcare System. Study 3: Videoconferencing Between Ambulances and Physician Manned Rapid Response Vehicles, Effects on On-site Patient Treatment and Pattern of Referral
Brief Title: Videoconferencing Between Ambulances and Physician Manned Rapid Response Vehicles, Effects on On-site Patient Treatment and Patterns of Referral
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Central Denmark Region (Other)
Responsible Party: Principal Investigator, Nikolaj Raaber, MD, University of Aarhus
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRAA3
Record Dates: First submitted 2014-03-12; First posted 2014-03-21 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: All Acutely Ill or Injured Patients Receiving Care by Ambulance Personnel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Video consultation (Experimental): Patients in this arm receive video consultation from physician in doctor manned rapid response vehicle.
  Interventions: Device: iPad air with 4G/3G SIM card
- Telephone consultation (Active Comparator): Patients receiving prehospital care by ambulance personnel whom receive telephone consultation/supervision by physician in rapid response vehicle.
  Interventions: Device: iPad air with 4G/3G SIM card

INTERVENTIONS:
Device: iPad air with 4G/3G SIM card — iPad air with 4G/3G SIM card is used as device for videoconferencing. LifeSizeClearSea solution is used for videoconferencing.
  Video consultation
  Other Names: LifeSizeClearSea

SUMMARY:
Physician manned rapid response vehicles are a limited resource in the prehospital handling of acute patients.

In this study mobile videoconferencing between ambulances and the rapid response vehicles enables patient consultation at a distance. Video consultation between patient and the prehospital physician can take place when the patient is at home or in the ambulance.

The primary aim of this study is to examine the effect of video consultation between physician manned rapid response vehicles and patients receiving treatment by ambulance personnel on the number of patients receiving final treatment on-site in the pre-hospital setting

ELIGIBILITY:
Inclusion Criteria:

* All patients receiving prehospital care by ambulance personnel
* Must receive either telephone or video consultation by physician in rapid response vehicle

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2014-11 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients receiving final treatment on-site prehospitally | Final treatment is registered for the present consultation, expected assesment averagely within 1 hour. Expected to be presented up to 36 months after assessment

SECONDARY OUTCOMES:
Readmission | Within 3 days of primary contact. Will be assessed up to 24 months after primary contact. Expected to be presented up to 36 months after assessment.
  For all patients receiving consultation from physician manned rapid response vehicles the number of patients admitted to hospital within 3 days will assessed.
Change in site of referral | If destination for patient is changed during consultatation with physician it wille be assessed at the end of consultation, expected averagely to be within 1 hour after consultation, expected to presented up to 24 months after primary assessment
  If the department to receive the patient is changed during consultation between physician in rapid response vehicle and patient
Number of treatments delivered by ambulance personnel | The number of treatments delivered by ambulance personnel during consultation with physician in rapid response vehicle. Expected to be assessed averagely within 1 hour of consultation. Expected to be presented up 36 months after primary assessment

OTHER OUTCOMES:
Ambulance staff evaluation of usability of equipment | 1 day
  Is investigated by the use of survey
Physicians evaluation of equipment | 1 day
  Is investigated by the use of survey
Patient satisfaction | Within 3 weeks after receiving consultation
  Is investigated by telephone survey.

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaj Raaber, MD, Principal Investigator — Central Denmark Region; Erika Christensen, MD, medical director, Study Director — Central Denmark Region
Locations (2):
- Denmark (2):
  - Lægebilen, Hospitalsenheden Horsens, Horsens
  - Responce A/S, Horsens